CLINICAL TRIAL: NCT06049108
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-LY3871801 in Healthy Male Participants
Brief Title: A Study of Carbon-14-Labelled [14C] LY3871801 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18337; J3P-MC-FTAE (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-LY3871801 (Experimental): Single dose of [¹⁴C]-LY3871801 administered orally
  Interventions: Drug: [14C]-LY3871801

INTERVENTIONS:
Drug: [14C]-LY3871801 — Administered orally

SUMMARY:
The main purpose of this study is to evaluate how much of the study drug (LY3871801), administered as a single dose that has the radioactive substance 14C incorporated into it, passes from blood into urine, feces and expired air in healthy male participants. The study will also measure how much of the study drug gets into the bloodstream, how its broken down, and how long it takes the body to get rid of it. The study will last up to approximately 9 weeks including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are overtly healthy as determined by medical evaluation
* Have a body mass index of 18.5 to 32.0 kilograms per meter squared (kg/m²), inclusive
* Males who agree to use highly effective or effective methods of contraception

Exclusion Criteria:

* Have known allergies to LY3871801, related compounds, or any components of the formulation, or a history of significant atopy
* Have received or intend to receive any vaccination within 30 days prior to dosing until the follow-up phone call
* Have participated in a radiolabeled drug study, where exposures are known to the investigator or designee, within 4 months prior to check-in, or participated in a radiolabeled drug study, where exposures are not known to the investigator or designee, within 6 months prior to check-in

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Urinary Excretion of LY3871801 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Predose up to Day 7 post dose
  Urinary Excretion of LY3871801 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Fecal Excretion of LY3871801 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Predose up to Day 7 post dose
  Fecal Excretion of LY3871801 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Curve Versus Time From zero to Infinity (AUC [0-∞]) of [¹⁴C]-LY3871801 | Predose up to Day 7 post dose
  PK: AUC [0-∞] of [¹⁴C]-LY3871801
PK: AUC [0-∞] of Total Radioactivity in Plasma and Whole Blood | Predose up to Day 7 post dose
  PK: AUC [0-∞] of Total Radioactivity in Plasma and Whole Blood
PK: Maximum Concentration (Cmax) of [¹⁴C]-LY3871801 | Predose up to Day 7 post dose
  PK: Cmax of [¹⁴C]-LY3871801
PK: Cmax of Total Radioactivity | Predose up to Day 7 post dose
  PK: Cmax of Total Radioactivity
Total Radioactivity Recovered in Urine, Feces, and Expired Air | Predose up to Day 7 post dose
  Total Radioactivity Recovered in Urine, Feces, and Expired Air
Total Number of Metabolites of LY3871801 | Predose up to Day 7 post dose
  Total Number of Metabolites of LY3871801

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No